CLINICAL TRIAL: NCT01920854
Title: A Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study of Intravenously Administered SFP in Healthy Volunteers
Brief Title: A Single Ascending Dose Study of Soluble Ferric Pyrophosphate Administered Intravenously in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockwell Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RMTI-SFP-9
Record Dates: First submitted 2013-06-28; First posted 2013-08-12 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Kidney Failure, Chronic Therapy; Hemodialysis
Keywords: Soluble Ferric Pyrophosphate, Pharmacokinetics, Iron, Hemodialysis
MeSH Terms: conditions — Renal Insufficiency | interventions — spleen fibrinolytic proteinase (human)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Soluble Ferric Pyrophosphate (Experimental): Group/Cohort Designation: Ascending doses of SFP. Each subject will receive a defined dose of SFP IV administered under double-blind conditions. Pharmacokinetics of iron will be measured using a validated assay for iron and transferrin bound iron.
  Interventions: Drug: soluble ferric pyrophosphate
- Control (Placebo Comparator): Group/Cohort Designation: Each subject will receive placebo IV administered under double-blind conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: soluble ferric pyrophosphate
  Other Names: SFP
  Arms: Soluble Ferric Pyrophosphate
Drug: Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of fixed ascending doses of intravenously administered Soluble Ferric Pyrophosphate

DETAILED DESCRIPTION:
* A total of 48 healthy volunteers will be studied.
* Depending on the safety profile at completion of the highest dose cohort, an additional 2 cohorts of subjects may be studied.
* Doses of SFP may be modified, depending on the PK and safety findings at each dose level.
* Cohorts may be dropped for safety or tolerability after discussion with the sponsor.
* There will be 6 active and 2 placebo subjects in each study cohort.
* Subjects in Cohorts 1-3 will receive ascending doses of SFP by intravenous infusion over 4 hours.
* Subjects in Cohorts 4-6 will receive ascending doses of SFP by intravenous infusion over 12 hours.

All subjects will be confined in the CRC for 1 day prior to study drug administration and for 2 additional days for safety assessments and completion of test procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 inclusive at the time of consent. This inclusion criterion will only be assessed at the first screening visit.
2. Male or non-pregnant, non-lactating female who is at least 90 days post-partum.
3. Subject is willing to comply with any applicable contraceptive requirements of the protocol.
4. Satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination (PE), vital signs, electrocardiogram (ECG) and laboratory evaluation (hematology, biochemistry, urinalysis) as assessed by the Investigator.
5. An understanding, ability and willingness to fully comply with study procedures and restrictions.
6. Ability to provide written, personally signed and dated informed consent to participate in the study, in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guideline E6 and applicable regulations, before completing any study-related procedures.
7. Body Mass Index (BMI) between 20.0 and 32.0 kg/m² inclusive. This inclusion criterion will only be assessed at the first screening visit.
8. Subjects must agree to discontinue all iron preparations for 14 days prior to study drug administration.

Exclusion Criteria:

1. Current or recurrent disease (e.g. cardiovascular, renal, liver, gastro-intestinal, malignancy or other conditions) that could affect the action, absorption or disposition of the investigational product utilized in this study, or could affect clinical or laboratory assessments.
2. Hemoglobin < 11 g/dL or Hematocrit < 30%.
3. Serum iron concentration ≤ 70 µg/dL (male or female).
4. Current or relevant previous history of physical or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or study procedures.
5. Significant illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
6. Current use of any medication (including prescription, over the counter [OTC], herbal or homeopathic preparations) within 14 days of first dose of investigational product. Exceptions are hormonal replacement therapy, hormonal contraceptives, acetaminophen and non-steroidal anti-inflammatory drugs.
7. Known or suspected intolerance or hypersensitivity to iron containing product(s).
8. History of alcohol or other substance abuse within the last year.
9. A positive screen for cotinine, alcohol or drugs of abuse.
10. Male subjects who consume more than 21 units of alcohol per week or three units per day. Female subjects who consume more than 14 units of alcohol per week or two units per day. 1 alcohol unit =1 beer = 1 wine (5oz) = 1 liquor (1.5 oz.).
11. A history of a positive human immunodeficiency virus (HIV) antibody screen, Hepatitis B surface antigen (HBsAg) or Hepatitis C virus (HCV) antibody screen.
12. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g. gum, patch). Ex-users must report that they have stopped using tobacco for at least 30 days prior to receiving the first dose of investigational product.
13. Routine consumption of more than five units of caffeine per day or subjects who experience caffeine withdrawal headaches. One caffeine unit is contained in the following items: one 6-oz. cup of coffee, two 12-oz. cans of cola, one 12-oz. cup of tea, three 1-oz. chocolate bars.
14. Donation of blood or blood products (e.g., plasma or platelets) within 60 days prior to receiving the first dose of investigational product.
15. Use of another investigational product within 30 days prior to receiving the first dose of investigational product or active enrolment in another drug or vaccine clinical study.
16. Pregnancy or intention to become pregnant before completing all study drug treatment.
17. Current medical status that, in the investigators opinion, would preclude participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond D Pratt, MD FACP, Study Director — Rockwell Medical Inc
Locations (1):
- Kalamazoo, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohorts 1 - 6 Placebo: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohorts 1 - 6 Placebo received IV D5W infused over either 4 hours (Cohorts 1, 2, 3, 6) or 12 hours (Cohorts 4, 5).
- Cohort 1 SFP: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohort 1 SFP received 2.5 mg IV SFP infused over 4 hours.
- Cohort 2 SFP: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohort 2 SFP received 5.0 mg IV SFP infused over 4 hours.
- Cohort 3 SFP: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohort 3 SFP received 7.5 mg IV SFP infused over 4 hours.
- Cohort 4 SFP: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohort 4 SFP received 15 mg IV SFP infused over 12 hours.
- Cohort 5 SFP: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohort 5 SFP received 20 mg IV SFP infused over 12 hours.
- Cohort 6 SFP: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohort 6 SFP received 10 mg IV SFP infused over 4 hours.
Period: Overall Study
Arm/Group | Cohorts 1 - 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Started | 12 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 11 | 6 | 6 | 6 | 5 | 6 | 5
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1 - 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP | Total
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 4 | 3 | 4 | 5 | 1 | 23
  Male | 8 | 4 | 2 | 3 | 2 | 1 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 12 | 6 | 6 | 6 | 5 | 5 | 6 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 8
  White | 9 | 5 | 5 | 6 | 4 | 5 | 5 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 6 (Mean Total Serum Iron, Baseline Corrected)
Description: Serum iron for Cohorts 1-3, 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Serum iron for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: The PK Population was defined as all subjects receiving a dose of SFP or placebo who had sufficient post-dose blood samples taken to estimate PK parameters for serum iron endpoints. All 48 enrolled subjects were included in the PK Population.
Measure: Mean (Standard Deviation); unit: micrograms/dL
Groups:
- Cohorts 1 - 3, 6 Placebo: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohorts 1 - 3, 6 Placebo received IV D5W infused over 4 hours.
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
micrograms/dL
  t = 0 hrs | 18.87125 (19.08355) | 14.625 (13.54503) | 20.13333 (9.256061) | 14.806 (10.09701) | 31.73333 (17.07579)
  t = 0.5 hrs | 19.25243 (12.97435) | 22.075 (15.44849) | 33.21167 (16.22149) | 41.53333 (17.55844) | 58.65 (21.0115)
  t = 1 hr | 23.555 (16.79989) | 40.34 (14.2365) | 47.45 (19.26954) | 67.24 (29.08003) | 95.21667 (18.84658)
  t = 2 hrs | 32.54286 (32.58808) | 73.15 (62.48) | 88.28333 (22.29039) | 119.34 (46.55242) | 150.3333 (22.43806)
  t = 3 hrs | 41.3125 (31.5142) | 77.64 (25.54981) | 112.7333 (29.95721) | 173.4 (17.38678) | 210 (26.54807)
  t = 4 hrs | 43.75 (39.09914) | 82.76 (10.01489) | 143.4167 (33.93585) | 206 (37.76242) | 241.5 (25.6963)
  t = 4.5 hrs | 46.99 (33.692) | 94.38 (12.827) | 150.8 (39.0858) | 196.25 (46.29885) | 258.3333 (32.20973)
  t = 5 hrs | 50.74714 (39.71965) | 88.88 (30.95007) | 135.26 (40.90584) | 207.5 (41.23469) | 238.1667 (27.28675)
  t = 6 hrs | 46.3375 (32.43362) | 86.1 (23.73584) | 118.6 (40.09489) | 179.0833 (40.56158) | 214.5 (31.14322)
  t = 7.5 hrs | 26.27143 (25.89638) | 49.33333 (35.15774) | 81.35 (18.15717) | 131.45 (31.91825) | 170.8333 (27.63633)
  t = 8 hrs | 20.1875 (19.10194) | 40.91667 (32.76452) | 60.02833 (38.13224) | 118.25 (38.3246) | 148 (28.2772)
  t = 9 hrs | 7.852857 (25.84383) | 30.75 (51.07636) | 44.21667 (20.25452) | 79.96 (32.5411) | 122.6833 (21.64813)
  t = 10 hrs | -0.1875 (18.48079) | -2.76 (32.67052) | 24.02833 (19.2209) | 64.68333 (37.53566) | 81.01667 (25.26099)
  t = 12 hrs | -11.8538 (20.68082) | -30.9866 (23.72293) | -5.89333 (17.29701) | 23.21667 (42.48879) | 32.91667 (22.9566)
  t = 12.5 hrs | -11.7838 (24.1043) | -31.966 (22.61386) | -10.3888 (20.13357) | 15.26667 (27.3353) | 28.13333 (32.85319)
  t = 14 hrs | -14.525 (23.13773) | -38.3883 (18.17201) | -22.5 (13.67333) | 0.895 (27.98098) | -6.56617 (24.95741)
  t = 16 hrs | -23.0004 (26.67792) | -39.5 (15.30849) | -19.905 (17.7931) | -12.35 (31.50294) | -23.5 (28.53482)
  t = 20 hrs | -16.7163 (29.37565) | -43.8 (13.72461) | -23.655 (21.6553) | -11.0612 (15.55449) | -35.55 (22.41006)
  t = 24 hrs | 10.34714 (16.82299) | 11.7 (33.80067) | 6.542 (13.5174) | 2.05 (15.61893) | -11.655 (20.10851)
  t = 36 hrs | -4.24286 (15.34727) | -43.7666 (28.14838) | -9.72167 (20.08234) | -12.2612 (17.42613) | -27.3 (15.28005)
  t = 48 hrs | 21.73286 (19.95647) | 11.47783 (44.51915) | 21.82333 (19.21886) | 41.4 (50.85712) | 48.46 (18.48764)

2. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 4, 5 (Mean Total Serum Iron, Baseline Corrected)
Description: Serum iron for Cohorts 1-3 and 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Serum iron for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Groups:
- Cohorts 4 and 5 Placebo: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohorts 4 and 5 Placebo received IV D5W infused over 12 hours.
Arm/Group | Cohorts 4 and 5 Placebo | Cohort 4 SFP | Cohort 5 SFP
Number analyzed (Participants) | 4 | 6 | 6
micrograms/dL
  t = 0 hrs | 22.575 (8.144272) | 15.55 (11.59451) | 7.888333 (33.94121)
  t = 0.5 hrs | 21.7 (13.11602) | 26.25 (13.70631) | 29.97167 (33.57264)
  t = 1 hr | 23 (11.37629) | 49.46667 (12.52576) | 68.23333 (44.6479)
  t = 2 hrs | 24.9325 (17.2084) | 77.62 (17.82826) | 107.6333 (43.33413)
  t = 4 hrs | 41.16667 (32.85869) | 140.2 (19.84187) | 197.6667 (46.28031)
  t = 6 hrs | 42.975 (36.03807) | 168.8 (35.75891) | 232 (48.90808)
  t = 9 hrs | 17.6 (41.26835) | 167.2 (42.3757) | 228.8333 (44.96851)
  t = 12 hrs | 2.175 (29.20575) | 176 (43.28972) | 214.5 (49.31835)
  t = 12.5 hrs | -5.53333 (28.14255) | 141.3833 (49.73572) | 208.1667 (51.0232)
  t = 14 hrs | -2.9 (24.60732) | 116.7 (47.4452) | 161.9667 (46.50513)
  t = 16 hrs | -19.1667 (15.64811) | 38.18 (30.55899) | 92.43833 (56.28477)
  t = 18 hrs | -12.3 (13.66711) | 25.84 (37.53582) | 47.605 (37.80162)
  t = 20 hrs | -5.2889 (7.137707) | -6.06667 (31.71553) | -3.09 (29.31886)
  t = 24 hrs | 21.62233 (19.48729) | -10.2333 (35.97225) | -20.0617 (26.62087)
  t = 30 hrs | 31.485 (48.38732) | -30.225 (27.25856) | -25.6333 (29.99492)
  t = 36 hrs | -0.52333 (21.42192) | -23.15 (40.39885) | -34.6333 (41.33162)
  t = 48 hrs | 34.03333 (13.70632) | 36.02 (26.44139) | 19.95 (39.70616)

3. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 6 (Mean Transferrin-bound Iron, Baseline Corrected)
Description: Samples for transferrin-bound iron for Cohorts 1-3, 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for transferrin-bound iron for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
micrograms/dL
  t = 0 hrs | 15.81588 (15.29313) | 27.45 (10.6442) | 24.76667 (12.58438) | 18.03333 (13.6192) | 34.47833 (22.29513)
  t = 0.5 hrs | 16.12875 (16.956) | 36.86667 (8.992145) | 46.41667 (11.35067) | 48.3 (16.06275) | 62.93333 (20.16231)
  t = 1 hr | 24.04125 (23.55888) | 51.73333 (10.18797) | 70.8 (14.34489) | 81.31667 (21.66614) | 102.8 (22.60044)
  t = 2 hrs | 26.3875 (17.3591) | 69.25 (11.37853) | 112.55 (17.88449) | 142.9 (27.52417) | 166.6667 (22.00606)
  t = 3 hrs | 36.7375 (24.39203) | 96.06667 (17.22355) | 1148.3333 (26.3717) | 194.3333 (39.70222) | 223.6667 (21.58394)
  t = 4 hrs | 42.5375 (27.70637) | 111.4167 (21.85437) | 179.1667 (35.79618) | 229.8333 (58.21483) | 247.8333 (28.47045)
  t = 4.5 hrs | 46.3125 (26.86966) | 113 (10.55936) | 183.5 (37.35639) | 230.5 (54.47844) | 259.1667 (36.66833)
  t = 5 hrs | 47.8375 (31.67153) | 105.95 (21.48299) | 171.3333 (34.4248) | 240.6667 (42.41541) | 241.8333 (21.80291)
  t = 6 hrs | 39.7125 (23.02839) | 95.5 (21.20547) | 149 (31.89357) | 188.95 (53.37429) | 222.8333 (26.60388)
  t = 7.5 hrs | 21.84125 (16.90949) | 62.58333 (27.26891) | 95.25 (18.04658) | 158.2667 (63.67312) | 175.8333 (27.83822)
  t = 8 hrs | 16.7375 (14.66799) | 50.58333 (27.42418) | 84.1 (23.7459) | 125.1 (50.25754) | 154.1667 (30.0494)
  t = 9 hrs | 3.245 (9.291451) | 30.23833 (30.05141) | 52.21667 (17.32494) | 104.1883 (51.15559) | 125.35 (23.78098)
  t = 10 hrs | -5.4175 (8.513109) | 4.028333 (21.84233) | 25.38333 (18.08142) | 67.95 (42.27547) | 87.16667 (31.49366)
  t = 12 hrs | -18.8714 (17.95569) | -22.0445 (14.59163) | -7.33333 (19.53363) | 28.65 (22.83486) | 32.745 (29.99864)
  t = 12.5 hrs | -22.8429 (22.18268) | -27.4617 (12.8595) | -10.2667 (22.21894) | 15.68333 (19.74056) | 24.82833 (38.29261)
  t = 14 hrs | -25.4481 (27.93334) | -33.9617 (16.56204) | -14.85 (28.31902) | 3.167167 (13.43837) | -6.195 (29.40307)
  t = 16 hrs | -29.4667 (32.86135) | -35.8 (16.87637) | -23.4283 (26.12766) | -12.0333 (33.63212) | -28.2167 (30.50996)
  t = 20 hrs | -20.7163 (31.3054) | -27.7 (30.14558) | -24.7233 (22.46531) | -18.1717 (16.19425) | -40.4883 (27.31494)
  t = 24 hrs | 14.05 (14.51925) | 21.505 (37.16592) | 0.116667 (16.23887) | 7.605 (22.55452) | -16.455 (21.98194)
  t = 36 hrs | -15.6767 (31.81849) | -39.8117 (31.90823) | -16.6567 (16.39093) | -11.74 (14.89775) | -37.3 (14.24949)
  t = 48 hrs | 25.4875 (16.85459) | 26.68333 (51.62024) | 35.36667 (12.16251) | 40.945 (32.03071) | 42.94 (12.77861)

4. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 4, 5 (Mean Transferrin-bound Iron, Baseline Corrected)
Description: Samples for transferrin-bound iron for Cohorts 1-3 and 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for transferrin-bound iron for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 4 and 5 Placebo | Cohort 4 SFP | Cohort 5 SFP
Number analyzed (Participants) | 4 | 6 | 6
micrograms/dL
  t = 0 hrs | 26.675 (10.10095) | 17.13333 (13.10836) | 22.31167 (25.13075)
  t = 0.5 hrs | 24.6 (12.80989) | 32.36667 (14.44322) | 46.76667 (25.7235)
  t = 1 hr | 31.35 (14.11772) | 56.01667 (12.43309) | 80.48333 (26.35234)
  t = 2 hrs | 35.75 (16.21532) | 93.36667 (16.01058) | 136.3333 (27.94041)
  t = 4 hrs | 50.9 (26.83927) | 152 (14.02854) | 222.5 (41.28801)
  t = 6 hrs | 55 (38.45179) | 186.8 (27.12379) | 255.5 (51.20059)
  t = 9 hrs | 24.285 (43.9688) | 181.3333 (34.92659) | 254.5 (60.24201)
  t = 12 hrs | -0.975 (28.42761) | 178.5 (47.26415) | 236.8333 (62.58887)
  t = 12.5 hrs | -3.86667 (28.73436) | 157.6667 (47.00496) | 237.8333 (68.42051)
  t = 14 hrs | -7.03333 (19.74369) | 117.3333 (45.18808) | 180.65 (69.86598)
  t = 16 hrs | -12.1867 (10.43401) | 57.75 (41.30815) | 114.3117 (73.84014)
  t = 18 hrs | -11.52 (11.5913) | 17.705 (33.84819) | 58.51667 (63.66288)
  t = 20 hrs | -0.67667 (20.99592) | -8.81667 (25.93025) | 12.61167 (53.50657)
  t = 24 hrs | 30.39 (23.14673) | -12.0567 (25.6596) | -9.53833 (41.94388)
  t = 30 hrs | 26.44667 (41.6933) | -18.8283 (30.65685) | -22.9778 (23.78139)
  t = 36 hrs | -5.4 (27.97803) | -28.1672 (32.82391) | -28.35 (35.19118)
  t = 48 hrs | 40.46667 (15.25036) | 41.026 (34.08901) | 30.78333 (48.96756)

5. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 6 (Mean Absolute Transferrin Saturation, Calculated)
Description: Samples for transferrin saturation for Cohorts 1-3, 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for transferrin saturation for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percentage of saturation
  t = 0 hrs | 25.70875 (18.521548) | 41.85 (12.577559) | 27.466667 (13.091626) | 26.383333 (10.936986) | 39.066667 (10.129495)
  t = 0.5 hrs | 26.375 (19.6707) | 45.583333 (12.795533) | 34.5 (12.94805) | 35.716667 (11.168781) | 47.85 (10.774368)
  t = 1 hr | 29.4125 (23.073141) | 49.533333 (13.224019) | 41.266667 (14.069921) | 45.016667 (11.995902) | 58.583333 (11.177373)
  t = 2 hrs | 29.5625 (21.098337) | 56.15 (13.052624) | 54.75 (15.895377) | 63.05 (13.895719) | 79.45 (14.417039)
  t = 3 hrs | 32.1875 (21.176904) | 64.666667 (16.043898) | 65.866667 (17.335128) | 78.15 (14.831015) | 96.066667 (12.873176)
  t = 4 hrs | 33.9625 (22.445867) | 69.883333 (16.560002) | 75.233333 (19.819048) | 88.8 (11.348128) | 102.83333 (7.5210815)
  t = 4.5 hrs | 34.1 (21.703917) | 64.6 (12.73185) | 74.25 (20.471614) | 88.24 (13.994034) | 102.93333 (10.715721)
  t = 5 hrs | 34.825 (24.362251) | 66.8 (16.702934) | 70.983333 (19.212227) | 89.516667 (12.587679) | 98.716667 (9.4961922)
  t = 6 hrs | 32.75 (21.835816) | 64 (16.355427) | 64.116667 (18.901896) | 74.133333 (19.031938) | 93.966667 (11.727688)
  t = 7.5 hrs | 29.375 (24.115659) | 53.083333 (16.412973) | 49.316667 (16.104089) | 65.2 (18.721218) | 80.483333 (13.813532)
  t = 8 hrs | 25.38625 (17.277825) | 49.183333 (15.874182) | 44.9 (17.190579) | 56.15 (19.282298) | 74.316667 (15.067902)
  t = 9 hrs | 23.18875 (18.870984) | 41.866667 (14.993421) | 35.533333 (15.038972) | 50.483333 (18.139506) | 65.816667 (13.489613)
  t = 10 hrs | 19.4325 (13.439108) | 34.466667 (13.005794) | 27.416667 (13.433453) | 40.133333 (17.189842) | 55.366667 (15.617127)
  t = 12 hrs | 16.518571 (9.4347451) | 25.916667 (9.637306) | 17.828333 (11.615611) | 28.783333 (13.911925) | 39.866667 (13.873812)
  t = 12.5 hrs | 15.968571 (9.7540546) | 24.566667 (8.6832406) | 16.771667 (11.701778) | 25.618333 (12.537496) | 36.866667 (14.673196)
  t = 14 hrs | 15.332857 (7.8527208) | 22.483333 (8.5307483) | 15.301667 (8.8581091) | 21.486667 (10.91862) | 28.716667 (13.00514)
  t = 16 hrs | 13.305714 (3.6857693) | 23.366667 (10.372592) | 12.835 (6.5323617) | 15.85 (4.4440972) | 22.2 (12.467879)
  t = 20 hrs | 14.835 (4.4686303) | 25.916667 (10.491981) | 12.386667 (4.4342606) | 16.025 (7.9655351) | 18.633333 (10.414157)
  t = 24 hrs | 24.4125 (10.022038) | 40 (8.7824826) | 19 (5.8845561) | 22.733333 (8.7016474) | 24.483333 (8.0759932)
  t = 36 hrs | 16.454286 (5.1594536) | 19.883333 (5.2162886) | 14.198333 (6.6138655) | 17.441667 (9.7067696) | 18.213333 (5.4371561)
  t = 48 hrs | 27.55 (15.727683) | 40.533333 (14.972864) | 29.383333 (11.362291) | 31.766667 (17.181928) | 41.58 (8.2156558)

6. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 4, 5 (Mean Absolute Transferrin Saturation, Calculated)
Description: Samples for transferrin saturation for Cohorts 1-3 and 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for transferrin saturation for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of saturation
Arm/Group | Cohorts 4 and 5 Placebo | Cohort 4 SFP | Cohort 5 SFP
Number analyzed (Participants) | 4 | 6 | 6
percentage of saturation
  t = 0 hrs | 30.95 (3.2583227) | 26.5 (10.784062) | 32.45 (10.532379)
  t = 0.5 hrs | 31.55 (4.2930176) | 32.6 (11.667219) | 41.3 (11.031591)
  t = 1 hr | 32.875 (4.7422744) | 38.633333 (11.449658) | 50.283333 (10.526997)
  t = 2 hrs | 34.525 (5.4267086) | 50 (12.552928) | 67.266667 (13.599069)
  t = 4 hrs | 38.95 (7.485319) | 67.55 (12.12151) | 92.833333 (14.211498)
  t = 6 hrs | 40.625 (11.092452) | 73.56 (12.108179) | 108.86667 (16.846325)
  t = 9 hrs | 31.925 (12.673956) | 78.7 (16.428025) | 107.55 (6.8625797)
  t = 12 hrs | 23.7 (7.7948701) | 78.816667 (17.543935) | 104.9 (10.529008)
  t = 12.5 hrs | 21.766667 (6.7337459) | 71.483333 (20.245238) | 100.31667 (12.198429)
  t = 14 hrs | 20.333333 (3.6855574) | 57.733333 (15.467471) | 82.15 (15.394902)
  t = 16 hrs | 18.833333 (0.5507571) | 38.366667 (13.245628) | 61.3 (17.549473)
  t = 18 hrs | 18.766667 (1.5821926) | 26.5 (10.654201) | 43.433333 (14.76383)
  t = 20 hrs | 22.133333 (5.0895317) | 19.238333 (7.7310036) | 29.966667 (11.375178)
  t = 24 hrs | 30.766667 (4.5763887) | 17.683333 (4.5845029) | 22.783333 (7.0024043)
  t = 30 hrs | 30.266667 (11.83737) | 15.983333 (3.8012717) | 18.45 (5.9949145)
  t = 36 hrs | 20.7 (7.2297994) | 13.403333 (6.1446128) | 17.383333 (8.9302669)
  t = 48 hrs | 33.133333 (3.1817186) | 32.44 (17.400661) | 34.633333 (12.038383)

7. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 6 (Mean Total Iron Binding Capacity, Absolute)
Description: Samples for total iron binding capacity for Cohorts 1-3, 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for total iron binding capacity for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
micrograms/dL
  t = 0 hrs | 350 (44.2) | 318 (28.3) | 334 (23.8) | 352 (53.1) | 352 (35.9)
  t = 0.5 hrs | 344 (41.6) | 312 (27.3) | 328 (24.9) | 344 (54.5) | 348 (37.5)
  t = 1 hr | 345 (51.6) | 318 (29.5) | 334 (22.8) | 348 (53.9) | 352 (35.7)
  t = 2 hrs | 346 (45.6) | 312 (31.9) | 330 (29.9) | 347 (56.6) | 342 (36.6)
  t = 3 hrs | 348 (43) | 313 (28.5) | 329 (26.6) | 344 (52.8) | 342 (38.4)
  t = 4 hrs | 348 (41.1) | 312 (29.4) | 328 (23.4) | 340 (51.2) | 341 (37.4)
  t = 4.5 hrs | 359 (45.1) | 324 (35.7) | 339 (22.3) | 337 (46.9) | 352 (35.5)
  t = 5 hrs | 358 (43.6) | 318 (27.6) | 338 (24.4) | 352 (42.6) | 350 (37.9)
  t = 6 hrs | 356 (44) | 315 (26) | 338 (24.8) | 356 (53.6) | 348 (37.8)
  t = 7.5 hrs | 347 (56.1) | 318 (27) | 332 (29.3) | 355 (52.8) | 348 (36.1)
  t = 8 hrs | 359 (38.6) | 319 (27.7) | 339 (25.2) | 356 (54.4) | 348 (34.6)
  t = 9 hrs | 348 (51.6) | 324 (27) | 338 (29.6) | 351 (47.2) | 349 (34.9)
  t = 10 hrs | 352 (41.4) | 317 (26.7) | 338 (28.8) | 355 (52.4) | 347 (34.6)
  t = 12 hrs | 351 (43) | 319 (26.3) | 333 (29.5) | 360 (53.5) | 344 (33.5)
  t = 12.5 hrs | 344 (52.7) | 316 (30.7) | 336 (23.5) | 351 (46.3) | 350 (25.8)
  t = 14 hrs | 340 (61.9) | 316 (31.1) | 335 (31.8) | 356 (48.4) | 344 (39.6)
  t = 16 hrs | 341 (41.1) | 304 (46.8) | 327 (27.1) | 353 (27.5) | 344 (36.9)
  t = 20 hrs | 342 (48.8) | 301 (40.8) | 326 (23.4) | 350 (52.3) | 338 (32.4)
  t = 24 hrs | 355 (43.4) | 314 (30.8) | 346 (22.6) | 362 (50) | 353 (35)
  t = 36 hrs | 362 (39.4) | 318 (24.8) | 344 (24.6) | 364 (50.4) | 357 (38.4)
  t = 48 hrs | 364 (43.2) | 320 (30.5) | 346 (19.3) | 370 (54.4) | 352 (36.3)

8. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 4, 5 (Mean Total Iron Binding Capacity, Absolute)
Description: Samples for total iron binding capacity for Cohorts 1-3 and 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for total iron binding capacity for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 4 and 5 Placebo | Cohort 4 SFP | Cohort 5 SFP
Number analyzed (Participants) | 4 | 6 | 6
micrograms/dL
  t = 0 hrs | 345 (22.3) | 346 (49.8) | 340 (41.1)
  t = 0.5 hrs | 332 (18.8) | 328 (41.8) | 328 (36.6)
  t = 1 hr | 340 (15.9) | 338 (42) | 336 (40.4)
  t = 2 hrs | 337 (17.6) | 336 (43.8) | 335 (36.6)
  t = 4 hrs | 338 (19.1) | 336 (42.4) | 335 (43.7)
  t = 6 hrs | 334 (22.9) | 338 (40.8) | 317 (41.3)
  t = 9 hrs | 330 (19.5) | 324 (37.8) | 318 (37.7)
  t = 12 hrs | 334 (33.3) | 319 (40.2) | 308 (35.1)
  t = 12.5 hrs | 333 (20.8) | 325 (37.1) | 323 (35.1)
  t = 14 hrs | 339 (19.3) | 328 (41.7) | 325 (31.8)
  t = 16 hrs | 338 (21.4) | 340 (37.8) | 325 (32.2)
  t = 18 hrs | 342 (13.9) | 337 (40.2) | 330 (34.3)
  t = 20 hrs | 337 (18.9) | 329 (40.4) | 325 (39)
  t = 24 hrs | 346 (31.2) | 344 (43.3) | 342 (39.4)
  t = 30 hrs | 344 (28.3) | 339 (42.2) | 350 (35.1)
  t = 36 hrs | 346 (33.7) | 344 (46.4) | 345 (35.4)
  t = 48 hrs | 352 (20.8) | 337 (42.6) | 343 (38.8)

9. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 6 (Mean Non-transferrin Bound Iron, Baseline Corrected)
Description: Samples for non-transferrin bound iron for Cohorts 1-3, 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for non-transferrin bound iron for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
micrograms/dL
  t = 0 hrs | 2.98 (7.07) | -5.44 (5.35) | -4.66 (6.42) | -4.74 (7.01) | -1.42 (5.22)
  t = 0.5 hrs | 5.93 (11.5) | -7.54 (8.74) | -13.2 (9.7) | -7.65 (21.8) | -4.92 (6.33)
  t = 1 hr | -0.554 (11.6) | -2.51 (10.1) | -23.4 (9) | -13.9 (35.8) | -7.54 (3.74)
  t = 2 hrs | 5.07 (19.6) | 12 (53.5) | -24.5 (11.9) | -26.9 (29.5) | -13.8 (6.34)
  t = 3 hrs | 4.5 (15.9) | -11.9 (10.3) | -35.6 (9.85) | -23.7 (30.1) | -9.69 (6.81)
  t = 4 hrs | 1.17 (12.6) | -13.2 (19.8) | -35.7 (16.4) | -24.3 (23.5) | -6.96 (5.75)
  t = 4.5 hrs | 0.0952 (13.2) | -9.79 (26.5) | -32.9 (16.5) | -27 (22) | 0.744 (13.3)
  t = 5 hrs | 1.01 (15.4) | -10.7 (11.5) | -32.7 (15) | -34 (19.7) | -2.92 (15.3)
  t = 6 hrs | 6.55 (20.1) | -10.1 (11.3) | -30.4 (13.4) | -11 (28) | -7.16 (13.5)
  t = 7.5 hrs | 3.3 (14.5) | -6.01 (10.1) | -13.9 (13.6) | -27.4 (44.4) | -5.09 (16.5)
  t = 8 hrs | 3.37 (10.6) | -2.43 (9.75) | -24 (20.1) | -7.72 (25.1) | -5.74 (11.1)
  t = 9 hrs | 6.31 (20.8) | 7.69 (26.8) | -8.02 (7.3) | -27 (36) | -2.44 (16.2)
  t = 10 hrs | 5.16 (12.8) | 1.51 (6.03) | -1.37 (4.46) | -4.22 (31.2) | -5.56 (11.3)
  t = 12 hrs | 9.52 (14.9) | -3.11 (9.14) | 1.43 (5.26) | -6.32 (42.9) | -0.472 (16.2)
  t = 12.5 hrs | 12.7 (21.2) | 1.17 (9.66) | -0.139 (6.84) | -1.3 (30.4) | 2.66 (11.1)
  t = 14 hrs | 11 (12.8) | 2.82 (12.6) | -3.44 (17.9) | -3.15 (28.3) | -1.01 (6.73)
  t = 16 hrs | 6.32 (11.1) | 4.85 (12.7) | 3.51 (10.3) | -1.2 (32.5) | 4.08 (10.7)
  t = 20 hrs | 3.92 (9.3) | 0.353 (22.2) | 1.06 (6.27) | 6.22 (25.3) | 4.29 (6.91)
  t = 24 hrs | -3.37 (4.87) | -6.39 (12.5) | 5.47 (5.98) | -6.43 (31.1) | 4.16 (9.23)
  t = 36 hrs | 2.97 (10) | 1.51 (15.2) | 6.93 (5.2) | -1.4 (23.6) | 9.36 (8.63)
  t = 48 hrs | -6.73 (14.6) | -7.56 (11.7) | -13.6 (19.7) | -1.65 (24.3) | 4.74 (14.3)

10. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 4, 5 (Mean Non-transferrin Bound Iron, Baseline Corrected)
Description: Samples for non-transferrin bound iron for Cohorts 1-3 and 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for non-transferrin bound iron for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 4 and 5 Placebo | Cohort 4 SFP | Cohort 5 SFP
Number analyzed (Participants) | 4 | 6 | 6
micrograms/dL
  t = 0 hrs | -4.08 (2.22) | -1.58 (2.45) | -13.9 (25.8)
  t = 0.5 hrs | -7.44 (8.71) | -5.95 (7.54) | -14.8 (26.7)
  t = 1 hr | -6.63 (4.35) | -5.93 (8.93) | -9.99 (38.2)
  t = 2 hrs | -10.4 (7.52) | -12.9 (23.4) | -20.7 (28.1)
  t = 4 hrs | -6.57 (4.26) | -10.1 (8.65) | -17.6 (28.7)
  t = 6 hrs | -10.8 (12.3) | -15.8 (16.4) | -18.1 (28.6)
  t = 9 hrs | -6.53 (13.2) | -10.1 (18.3) | -19.8 (28.2)
  t = 12 hrs | 3.17 (2.29) | -11.7 (12.8) | -18.4 (22.4)
  t = 12.5 hrs | -1.63 (1.54) | -16.3 (15.5) | -20.2 (28.3)
  t = 14 hrs | 0.0167 (1.39) | -3.38 (7.01) | -14.2 (33.5)
  t = 16 hrs | -6.97 (13.6) | -6.93 (9.07) | -17.9 (29.5)
  t = 18 hrs | -0.767 (9.7) | 1.81 (8.29) | -8.14 (28)
  t = 20 hrs | -4.6 (14.9) | 2.75 (8.15) | -14.4 (31)
  t = 24 hrs | -8.63 (8.31) | 1.83 (16.3) | -10.8 (27.5)
  t = 30 hrs | -3.68 (3.09) | 1.22 (9.34) | -2.87 (35.6)
  t = 36 hrs | 4.9 (9.01) | 5.32 (20.5) | -6.44 (29.2)
  t = 48 hrs | -4.63 (1.7) | -4.03 (22.1) | -8.46 (36.1)

11. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 6 (Mean Unbound Iron Binding Capacity, Baseline Corrected)
Description: Samples for unbound iron binding capacity for Cohorts 1-3, 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for unbound iron binding capacity for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
micrograms/dL
  t = 0 hrs | -15.7 (16.3) | -27 (9.55) | -22.9 (10.7) | -17.9 (13.9) | -37.4 (24)
  t = 0.5 hrs | -22.4 (19.4) | -41.5 (7.97) | -50.2 (10.7) | -56.8 (17.3) | -70.7 (23.8)
  t = 1 hr | -29.1 (34.7) | -51.1 (9.91) | -68.7 (10.6) | -85.9 (19.2) | -106 (22.6)
  t = 2 hrs | -30.3 (24.2) | -74.1 (10.9) | -115 (22.9) | -148 (25.9) | -179 (25.1)
  t = 3 hrs | -38.9 (26.7) | -100 (21.4) | -152 (26.2) | -201 (39.2) | -229 (30.6)
  t = 4 hrs | -44.8 (31.2) | -117 (22.6) | -182 (36.1) | -242 (58.8) | -246 (29.4)
  t = 4.5 hrs | -37.9 (33.2) | -103 (10.6) | -175 (34.5) | -222 (59.4) | -243 (30.8)
  t = 5 hrs | -39.9 (37.8) | -105 (25.5) | -166 (35.9) | -237 (60.6) | -239 (30.5)
  t = 6 hrs | -34.5 (29.7) | -97.3 (25.8) | -143 (31.4) | -185 (50.9) | -228 (33.5)
  t = 7.5 hrs | -25.1 (35.4) | -61.8 (28.7) | -95.3 (26.9) | -156 (68.9) | -183 (32.3)
  t = 8 hrs | -8.54 (15.5) | -48.9 (26.6) | -77.4 (26.2) | -121 (52.5) | -161 (34.8)
  t = 9 hrs | -5.54 (23.6) | -23.6 (22.9) | -46.5 (25.5) | -106 (56.4) | -132 (29.7)
  t = 10 hrs | 7 (12) | -3.71 (18.1) | -20 (23.6) | -65.7 (50.1) | -95.5 (34.9)
  t = 12 hrs | 19.4 (10.5) | 24.4 (13.7) | 8.56 (26.4) | -21.5 (33.7) | -43.7 (32)
  t = 12.5 hrs | 17.1 (10.6) | 26 (13.6) | 14 (32) | -16.7 (33.7) | -30.6 (34.4)
  t = 14 hrs | 16 (8.71) | 32.8 (11.5) | 17.7 (37.1) | 0.667 (20) | -5.4 (34.1)
  t = 16 hrs | 21 (24.1) | 22.5 (21.5) | 18.5 (30.1) | 10.8 (10.6) | 16.5 (33.1)
  t = 20 hrs | 11.8 (19.4) | 11.9 (28.5) | 19 (25.4) | 15.3 (15.5) | 23.1 (26.3)
  t = 24 hrs | -9.1 (13.8) | -24.7 (32.2) | 13.8 (22.8) | 1.57 (23) | 14 (16.5)
  t = 36 hrs | 28.1 (28.6) | 41.1 (30.1) | 28.6 (19.5) | 23.1 (15.1) | 38.7 (21.1)
  t = 48 hrs | -12.2 (25.3) | -23.4 (46.3) | -21.1 (16) | -23.8 (38.3) | -44.4 (18.4)

12. Primary Outcome: Pharmacokinetics of Iron From Soluble Ferric Pyrophosphate: Cohorts 4, 5 (Mean Unbound Iron Binding Capacity, Baseline Corrected)
Description: Samples for unbound iron binding capacity for Cohorts 1-3 and 6 will be collected at 0, 0.5,1, 2, 3, 4, 4.5, 5, 6, 7, 7.5, 8, 9,10, 12,12.5 14, 16, 20, 24,36, and 48 hours. Samples for unbound iron binding capacity for Cohorts 4 and 5 will be collected at 0, 0.5,1, 2, 4, 6, 9, 12,12.5, 14,16,18,20, 24, 30, 36, and 48 hours.
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL
Arm/Group | Cohorts 4 and 5 Placebo | Cohort 4 SFP | Cohort 5 SFP
Number analyzed (Participants) | 4 | 6 | 6
micrograms/dL
  t = 0 hrs | -19.7 (8.82) | -12.4 (17.6) | -19.4 (29.5)
  t = 0.5 hrs | -30.4 (11.6) | -46.5 (9.79) | -56.3 (29.7)
  t = 1 hr | -29.7 (16.2) | -59.8 (8.85) | -81.3 (29.2)
  t = 2 hrs | -37.1 (19.2) | -99.2 (14) | -138 (32.9)
  t = 4 hrs | -51.2 (25.8) | -158 (21.6) | -216 (27.9)
  t = 6 hrs | -58.7 (41.6) | -189 (38.5) | -247 (37.5)
  t = 9 hrs | -32.4 (46.3) | -199 (41.6) | -246 (44.2)
  t = 12 hrs | -3.59 (30.8) | -201 (51.9) | -241 (51.8)
  t = 12.5 hrs | -1.21 (29.8) | -174 (66.1) | -236 (60.7)
  t = 14 hrs | 8.29 (17.2) | -131 (52.9) | -193 (76.1)
  t = 16 hrs | 11.8 (11.2) | -59.7 (58.2) | -126 (76.4)
  t = 18 hrs | 15.4 (20.3) | -22.3 (44.6) | -65.7 (65.6)
  t = 20 hrs | -0.0778 (30.5) | -3.63 (33.6) | -24.7 (52.8)
  t = 24 hrs | -22.8 (33.3) | 14.6 (24.6) | 14.3 (49.4)
  t = 30 hrs | -20.9 (53.3) | 15.9 (35.5) | 35.8 (28.1)
  t = 36 hrs | 13.7 (39.4) | 30.1 (37.7) | 36.6 (34.6)
  t = 48 hrs | -26.2 (25.3) | -35.8 (36.2) | -24.5 (54.8)

13. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean AUC [Area Under the Curve] 0 - 12, Mean AUC 0 - 4, Mean AUC Last)
Description: Samples for three area under the curve (AUC) calculations (AUC 0-12, AUC 0 - 4, and AUC last) were collected for all Cohorts (both SFP and placebo).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*microgram/dL
Groups:
- Cohorts 1 - 3, 6 Placebo: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohorts 1 -3, 6 Placebo received IV D5W infused over 4 hours.
- Cohorts 4, 5 Placebo: A total of 48 subjects were studied in 6 sequential cohorts (8 subjects per group, randomized as 6 active and 2 placebo). Cohorts 1, 2, 3, and 6 received ascending doses of test article over 4-hour infusions. Cohorts 4 and 5 received ascending doses of test article over 12-hour infusions. Cohorts 4, 5 Placebo received IV D5W infused over 12 hours.
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohorts 4, 5 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 4 | 6 | 6 | 6 | 6 | 6 | 6
h*microgram/dL
  AUC 0 - 12 | 289 (235) | 334 (412) | 546 (312) | 890 (258) | 1420 (316) | 1590 (336) | 2210 (402) | 1770 (222)
  AUC 0 - 4 | 126 (103) | 107 (68.8) | 235 (104) | 329 (84.8) | 471 (97.7) | 305 (56) | 426 (151) | 590 (76.7)
  AUC last | 340 (206) | 277 (409) | 579 (265) | 903 (261) | 1460 (340) | 2070 (639) | 3000 (677) | 1820 (263)

14. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean AUC [Area Under the Curve] Inf)
Description: Samples for area under the curve from time-zero extrapolated to infinity (AUC inf) calculations were collected for all Cohorts (just those subjects that received SFP).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*microgram/dL
Arm/Group | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
h*microgram/dL | 675 (270) | 1010 (190) | 1650 (172) | 2340 (565) | 3150 (657) | 1840 (263)

15. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean CL [Clearance])
Description: Samples for Clearance (CL) calculations were collected for all Cohorts (just those subjects that received SFP).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dL/hour
Arm/Group | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
dL/hour | 4.06 (1.2) | 5.11 (0.99) | 4.59 (0.464) | 6.72 (1.63) | 6.61 (1.5) | 5.56 (0.938)

16. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (C Max)
Description: Samples maximal baseline corrected concentration of iron (Cmax) calculations were collected for all Cohorts (both SFP and placebo).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/dL
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohorts 4, 5 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 8 | 4 | 6 | 6 | 6 | 6 | 6 | 6
microgram/dL | 62.6 (32.4) | 44.3 (34.8) | 113 (44.5) | 151 (33.9) | 228 (19.7) | 177 (38.2) | 251 (51.7) | 261 (30.3)

17. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Tmax)
Description: Samples for observed time to reach maximum iron concentration (Tmax) calculations were collected for all Cohorts (both SFP and placebo).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Cohorts 1 - 3, 6 Placebo | Cohorts 4, 5 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 12 | 4 | 6 | 6 | 6 | 6 | 6 | 6
hours | 4.5 [0.5 to 6] | 6 [4 to 6] | 4.5 [2 to 9] | 4.5 [4 to 4.5] | 4.75 [4 to 6] | 7.5 [6 to 12] | 6 [4 to 12.1] | 4.5 [4 to 4.5]

18. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean Cmax/Dose)
Description: Samples for the dose-normalized maximal baseline corrected concentration of iron (Cmax/dose) calculations were collected for all Cohorts (just those subjects that received SFP).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrograms/dL/mg
Arm/Group | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
micrograms/dL/mg | 45.3 (17.8) | 30.2 (6.78) | 30.4 (2.63) | 11.8 (2.55) | 12.5 (2.59) | 26.1 (3.03)

19. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean Lambda z)
Description: Samples for terminal phase rate constant (lambda z) calculations were collected for all Cohorts (just those subjects that received SFP).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
1/hour | 0.544 (0.0788) | 0.668 (0.281) | 0.711 (0.423) | 0.475 (0.262) | 0.337 (0.114) | 0.917 (0.688)

20. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean Half Life: t 1/2)
Description: Samples for terminal phase half life (t 1/2) calculations were collected for all Cohorts (just those subjects that received SFP).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
hours | 1.3 (0.187) | 1.19 (0.476) | 1.29 (0.721) | 1.87 (1.08) | 2.21 (0.549) | 1.04 (0.505)

21. Secondary Outcome: Serum Iron Profile From Soluble Ferric Pyrophosphate: Cohorts 1, 2, 3, 4, 5, 6 (Mean Vz)
Description: Samples for volume of distribution in the terminal elimination phase (Vz) calculations were collected for all Cohorts (just those subjects that received SFP).
  There was no formal sample size calculation for this study; 48 subjects were enrolled and 48 subjects were analyzed to establish the PK profile of the serum iron from SFP. Study results were summarized by dose group, with descriptive statistics. No additional statistical testing was performed. No imputation of missing data was performed. No windowing of visits was performed.
Time Frame: 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dL
Arm/Group | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
dL | 7.65 (2.84) | 8.43 (2.94) | 8.59 (4.79) | 16.6 (6.33) | 20.8 (6.8) | 8.33 (4.05)

22. Primary Outcome: Baseline Transferrin Profile: Cohorts 1, 2, 3, 4, 5, 6
Description: The mean baseline transferrin will be calculated based on samples drawn just prior to infusion for all Cohorts (both SFP and placebo)
Time Frame: Baseline (1 day)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cohorts 1 - 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 6
mg/dL | 306.583 (35.1606) | 283.500 (29.9850) | 315.500 (40.7909) | 348.333 (59.9956) | 303.833 (47.2966) | 314.571 (52.6841) | 304.167 (53.2143)

ADVERSE EVENTS:
Arm/Group | Cohorts 1 - 6 Placebo | Cohort 1 SFP | Cohort 2 SFP | Cohort 3 SFP | Cohort 4 SFP | Cohort 5 SFP | Cohort 6 SFP
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/12 | 0/6 | 3/6 | 2/6 | 4/6 | 0/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohorts 1 - 6 Placebo (N=12) | Cohort 1 SFP (N=6) | Cohort 2 SFP (N=6) | Cohort 3 SFP (N=6) | Cohort 4 SFP (N=6) | Cohort 5 SFP (N=6) | Cohort 6 SFP (N=6)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
infusion site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vessel puncture site hemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
infusion site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less